CLINICAL TRIAL: NCT06158438
Title: Safety and Efficacy of the BTL-754 Device for Laser Skin Resurfacing Treatment of the Face
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTL-754_CTBG100
Record Dates: First submitted 2023-11-28; First posted 2023-12-06 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Wrinkle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (1):
- BTL-754-4 Treatment (Experimental): Treatment with BTL-754 device with the applicator BTL-754-4 for reduction of facial wrinkles.
  Interventions: Device: BTL-754-4 Treatment

INTERVENTIONS:
Device: BTL-754-4 Treatment — Treatment with the BTL-754 device with the BTL-754-4 applicator for reduction of facial wrinkles.

SUMMARY:
This study will evaluate the clinical safety and the performance of the BTL-754 device (equipped with the 754-4 applicator) for reduction of facial wrinkles by the means of laser skin resurfacing treatment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects over 22 years of age seeking treatment for reduction of wrinkles.
* Presence of clearly visible wrinkles in the treated area when the face is relaxed as deemed appropriate by the Investigator.
* Subjects are willing to have polycarbonate eye shields placed for study treatment.
* Subjects should be able to understand the investigative nature of the treatment, the possible benefits and side effects, and must sign the Informed Consent Form.
* Subjects are willing to maintain the usual skin care regimen during study participation with the exception when protocol specified ointments, moisturizers, and cleansers are required during the healing stage. Sunblock is required throughout the subject's participation in the study.
* Subjects are willing to abstain from other facial cosmetic procedures during the study; examples include, but are not limited to: laser or chemical resurfacing, dermabrasion, neuromodulator and/or filler injections, aesthetic facial surgery, etc.
* Subjects are willing and able to comply with protocol requirements, including obtaining study-required digital photographs and assessments, post-care instructions, and returning for follow-up visits.
* Women of childbearing potential are required to use birth control measures.

Exclusion Criteria:

* Intolerance to anesthetic based agents
* Infectious disease
* Connective tissue disease
* Propensity for keloid formations
* Immunocompromised or compromised healing
* Use of long-standing systemic steroids (e.g. Prednisone, Dexamethasone)
* Pregnant, planning to become pregnant, or breast feeding during the study
* Use of isotretinoin (e.g. Accutane, Sotret, Claravis, Amnesteem) within the past year
* Medical condition that may affect wound healing
* Any unstable medical or psychiatric conditions
* Major systemic diseases - e.g. uncontrolled Diabetes mellitus
* Photosensitivity, medications affecting sensitivity to light
* Corticosteroids or injections of the treated area within the last 90 days, long-term corticosteroids use
* Electronic implants (such as cardiac pacemakers, defibrillators and neurostimulators)
* Blepharoplasty (in case of eyelid treatment)
* Anticoagulant therapy, bleeding disorders
* Application within 4 to 6 months after radiotherapy
* Known or suspected malignancy, history of cancer or any type of malignancy
* Febrile conditions, serious illness, chronic infection
* Epilepsy
* Deep vein thrombosis
* Subject has had concurrent therapy that, in the investigator's opinion, would interfere with the evaluation of the safety and effectiveness of the study treatment method.
* Subject is enrolled in another investigational (drug or device) clinical trial or has participated in any other investigational study within 30 days prior to consent that can interfere with this study's assessments as per investigator's discretion.
* Subject has undergone a facelift procedure, IPL, laser, microneedling, chemical peels, dermal fillers, BOTOX® or other toxins within 6 months prior to the screening visit.
* Tattoo(s) or permanent make-up in the intended treatment area.
* Subject has used, within 30 days prior to screening or plans to use during study participation, Accutane, Retinol, or any medication that can cause dermal hypersensitivity.
* Any other disease or condition at the investigator discretion that may pose risk to the patient or compromise the study.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2023-11-16 (Actual); Primary Completion 2024-06-07 (Actual); Study Completion 2024-08-19 (Actual)

PRIMARY OUTCOMES:
Assess reduction of wrinkle severity according to the Fitzpatrick Wrinkle and Elastosis Scale | 5 months
  The primary efficacy outcome measure is a statistically significant reduction of at least 1.0 score in the average score of Fitzpatrick Wrinkle and Elastosis Scale score according to at least 2 out of 3 blinded dermatologists at 3-months follow-up compared to baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for specialized medical care - Individual dermatological practice Dr. Mariya Genova, Plovdiv, Plovdiv, Bulgaria

IPD SHARING:
Plan to Share IPD: No